CLINICAL TRIAL: NCT00176566
Title: A Phase II Trial to Assess the Effects of Green Tea in Oral Leukoplakia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Transitioned into a national study through ECOG
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Susan Goodin, Pharm.D., The Cancer Institute of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 4383; CINJ#120301
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Oral Leukoplakia
Keywords: oral leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Lozenge Intake — of green tea lozenges weighing 6 grams each, containing 0.45 grams of green tea solids eight (8) times daily for 12 weeks to patients with oral leukoplakia compared to the administration of a lozenge that does not contain green tea (i.e. a placebo lozenge).

SUMMARY:
You have been asked to participate in this research study because you have or may have oral leukoplakia. Oral leukoplakia is described as a white patch or plaque on the oral mucosa (mouth) that will not rub off and cannot be removed by scraping, reversed by elimination of obvious irritants (things that cause redness and/or swelling) such as dentures (artificial replacment for missing teeth), or lesions as described that are diagnosed by your dentist.

DETAILED DESCRIPTION:
Since oral leukoplakia may precede the development of cancer, using agents that may prevent cancer, called chemoprevention, may be useful. The purpose of this study is to determine whether taking a green tea preparation may have effects on your leukoplakia. It is hoped that these effects may reduce the subsequent risk of cancer in or around the area of leukoplakia. To assess for these effects, samples of the lining of your mouth will be obtained, and they will be analyzed looking for certain features (biomarkers).

ELIGIBILITY:
* Patients with oral leukoplakia without evidence of active infections in the mouth will be invited to participate in this study.
* Patients must currently consume no more than 3 cups of tea a day,
* not be taking large doses of vitamin A or its derivatives (more than 25,000 units), selenium, or beta-carotene.
* Additionally, patients must not participate in this study if they are allergic to caffeine, have GI ulcers, are pregnant, or have had previous invasive mouth cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of green tea lozenge versus placebo on the prevalence, size, and histologic severity of oral leukoplakia. | 3 years

SECONDARY OUTCOMES:
Additionally, we will correlate the changes in oral leukoplakia with levels of tea polyphenols in saliva and in biopsied lesions; DNA content in leukoplakia cells obtained from buccal scrapings; and proliferation index, apoptotic index, and expression of | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PharmD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- The Cancer Institute of New Jersey, New Brunswick, New Jersey, United States